CLINICAL TRIAL: NCT01609062
Title: A Randomized, Double-Blind, Pilot Study of the Safety and Physiological Effects of Two Doses of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Brief Title: Safety and Exercise Study of Two Doses of BMN 110 for Morquio A Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOR-008
Record Dates: First submitted 2012-05-24; First posted 2012-05-31 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Mucopolysaccharidosis IVA; Morquio A Syndrome; MPS IVA
Keywords: Mucopolysaccharidosis IVA Type A; MPS IVA Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT; MOR-008; CPET; MST; muscle strength test; physiological effect
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — GALNS protein, human; Chondroitinases and Chondroitin Lyases; Galns protein, mouse; Sulfatases; Enzyme Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMN 110 Weekly at 2.0 mg/kg/week (Experimental)
  Interventions: Drug: BMN 110
- BMN 110 Weekly at 4.0 mg/kg/week (Experimental)
  Interventions: Drug: BMN 110

INTERVENTIONS:
Drug: BMN 110 — Weekly IV infusions of BMN 110 at 2.0 mg/kg/week over a period of approximately 4 hours per infusion for up to 192 weeks.
  Other Names: N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT; elosulfase alfa
  Arms: BMN 110 Weekly at 2.0 mg/kg/week
Drug: BMN 110 — Weekly IV infusions of BMN 110 at 4.0 mg/kg/week over a period of approximately 4 hours per infusion for 27 weeks, and will eventually transition to 2.0 mg/kg/week for up to an additional 166 weeks.
  Other Names: N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT; elosulfase alfa
  Arms: BMN 110 Weekly at 4.0 mg/kg/week

SUMMARY:
The primary objective of this study was to evaluate the safety of a 2.0 mg/kg/week and a 4.0 mg/kg/week of BMN 110 in patients with Morquio A syndrome for up to 196 weeks. Secondary objectives were to investigate the effect of the two doses on exercise capacity for up to 196 weeks. In addition, the pharmacokinetic (PK) parameters of both doses of BMN 110 was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written, signed informed consent (or patient's legally authorized representative) after the nature of the study has been explained and prior to performance of any research- related procedure. Also, patients who do not meet country and local age requirements for informed consent must be willing and able to provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to performance of any research-related procedure.
* Has documented clinical diagnosis of Morquio A Syndrome (MPS IVA) based on clinical signs and symptoms of MPS IVA and documented reduced fibroblast or leukocyte N-acetylgalactosamine-6-sulfatase (GALNS) enzyme activity or genetic testing confirming diagnosis of MPS IVA.
* Is at least 7 years of age
* Is able to walk ≥ 200 meters as assessed by the 6-minute Walk Test (6MWT)
* If sexually active, is willing to use an acceptable method of contraception while participating in the study
* If female of childbearing potential, must have a negative pregnancy test at the Screening Visit and be willing to have additional pregnancy tests during the study
* Is willing and able to perform all study procedures, including cardiopulmonary exercise testing (CPET)

Exclusion Criteria:

* Inability to perform an exercise test due to limited mobility
* Body weight greater than 95 kg at Screening
* Severe, untreated sleep apnea as measured during Screening with a home sleep testing device
* Patients with a history of, or current condition of sleep apnea or sleep disordered breathing under adequate treatment may be enrolled if approved by the medical monitor.
* Requirement for supplemental oxygen
* Use of ventilator assistance in the 3 months prior to study entry
* Use of positive airway pressure (continuous positive airway pressure, CPAP, or bilevel airway pressure) for treatment of sleep apnea or sleep disordered breathing is allowed if settings have been stable for at least 1 month prior to study entry, and is approved by the medical monitor.
* Has a concurrent disease or condition, including but not limited to, symptomatic cervical spine instability, clinically significant spinal cord compression, or severe cardiac disease that would interfere with study participation, or pose a safety risk, as determined by the Investigator
* Has previous hematopoietic stem cell transplant (HSCT)
* Has received previous treatment with BMN 110
* Has a known hypersensitivity to BMN 110 or its excipients
* Has had major surgery within 3 months prior to study entry or is planning to have a major surgery during the duration of the study
* Use of any other investigational product (IP) or investigational medical device within 30 days prior to the beginning of the Screening Period or requires any investigational agent prior to completion of all scheduled study assessments
* Is pregnant or breastfeeding during the Screening Period or planning to become pregnant (self or partner) at any time during the study
* Has a concurrent disease or condition that may interfere with study participation or safety, and/or ability to perform study procedures as determined by the Investigator
* Has any condition that, in the view of the Investigator, poses a safety risk to the patient
* Has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Shaywitz, MD PhD, Study Director — BioMarin Pharmaceutical
Locations (11):
- United States (4):
  - Oakland, California
  - Chicago, Illinois
  - New York, New York
  - Houston, Texas
- Canada (4):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrook, Quebec
- Hamburg, Germany
- United Kingdom (2):
  - Belfast, Northern Ireland
  - Manchester

REFERENCES:
- [Derived] Berger KI, Burton BK, Lewis GD, Tarnopolsky M, Harmatz PR, Mitchell JJ, Muschol N, Jones SA, Sutton VR, Pastores GM, Lau H, Sparkes R, Shaywitz AJ. Cardiopulmonary Exercise Testing Reflects Improved Exercise Capacity in Response to Treatment in Morquio A Patients: Results of a 52-Week Pilot Study of Two Different Doses of Elosulfase Alfa. JIMD Rep. 2018;42:9-17. doi: 10.1007/8904_2017_70. Epub 2017 Nov 21. PMID 29159458

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 110 Weekly at 2.0 mg/kg/Week: BMN 110: Weekly IV infusions of BMN 110 at 2.0 mg/kg/week over a period of approximately 4 hours per infusion in the primary phase.
- BMN 110 Weekly at 4.0 mg/kg/Week: BMN 110: Weekly IV infusions of BMN 110 at 4.0 mg/kg/week over a period of approximately 4 hours per infusion in the primary phase.
Period: Primary Phase
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week
Started | 15 | 10
Completed | 15 | 10
Not Completed | 0 | 0
Period: Extension Phase
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week
Started | 15 | 10
Completed | 0 | 0 (EAP = Expanded Access Program)
Not Completed | 15 | 10
Not completed — Terminated by Sponsor | 14 | 9
Not completed — Discontinued drug and then was pregnant | 1 | 0
Not completed — Anticipated surgery & transition to EAP | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (9.32) | 12.0 (3.16) | 13.7 (7.52)
Age, Customized [Number; unit: participants]
  7 to 11 years | 9 | 5 | 14
  12 to 18 years | 3 | 5 | 8
  >=19 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 9 | 23
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 1 | 6
  Germany | 0 | 3 | 3
  United Kingdom | 1 | 1 | 2
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation
Description: The primary objective of the study is to evaluate the safety of weekly infusions of BMN 110; the safety variables included Adverse Events (AEs).
  The primary outcome measure data is presented in more detail under the Adverse Events section.
Time Frame: Entire Study Period, up to 192 weeks or ETV (early termination visit)
Population: The primary outcome measure data is presented in more detail under the Adverse Events section.
Measure: Number; unit: participants
Groups:
- All Subjects: Both groups combined
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
participants
  Serious Adverse Events | 3 | 2 | 5
  Other (Not Including Serious) Adverse Events | 15 | 10 | 25

2. Secondary Outcome: 6-minute Walk Test (6MWT)
Description: Change from baseline to Week 12, 24, and 52 as measured in distance walked (meters) in 6MWT.
Time Frame: Baseline, Week 12, 24, and 52
Population: Modified Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
meters
  Week 12 | 14.7 (30.90) | -8.9 (83.52) | 5.3 (57.55)
  Week 24 | -13.0 (54.12) | 0.1 (34.70) | -7.8 (46.94)
  Week 52 | 9.0 (48.41) | 31.8 (54.56) | 18.5 (51.19)

3. Secondary Outcome: 3-minute Stair Climb Test (3MSCT)
Description: Change from baseline to Week 12, 24, and 52 as measured in speed (stairs/min) in 3MSCT.
Time Frame: Baseline, Week 12, 24, and 52
Population: Modified Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: stairs/min
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
stairs/min
  Week 12 | -3.7 (13.16) | 1.7 (11.28) | -1.5 (12.49)
  Week 24 | -2.2 (11.01) | 12.5 (15.26) | 3.9 (14.65)
  Week 52 | -4.4 (9.82) | 10.0 (16.88) | 1.3 (14.66)

4. Secondary Outcome: Respiratory Function Test (MVV and FVC)
Description: Respiratory Function was assessed by spirometry in accordance with American Thoracic Society standards.
  Percent change from baseline to Week 12, 24, and 52 as measured by Maximum Voluntary Ventilation (MVV, L/min) Percent change from baseline to Week 12, 24, and 52 as measured by Forced Vital Capacity (FVC, L)
Time Frame: Baseline, Week 12, 24, and 52
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
Percent Change
  MVV Week 12 | 12.8 (21.77) | 32.4 (140.73) | 21.7 (94.00)
  MVV Week 24 | 8.8 (17.20) | -0.6 (27.00) | 4.3 (22.34)
  MVV Week 52 | 2.2 (41.24) | -17.8 (38.61) | -6.9 (40.43)
  FVC Week 12 | 1.7 (8.77) | 3.2 (10.63) | 2.3 (9.39)
  FVC Week 24 | 3.4 (9.01) | 13.0 (16.30) | 7.4 (13.16)
  FVC Week 52 | 4.8 (12.68) | 15.1 (15.94) | 8.9 (14.69)

5. Secondary Outcome: Normalized Urine Keratan Sulfate (uKS)
Description: Urinary KS was measured by a quantitative method and normalized using the sample urinary creatinine measurement.
  Percent change from baseline to Week 12, 24, and 52 in normalized urine keratan sulfate (ug/mg).
Time Frame: Baseline, Week 12, 24, and 52
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
Percent Change
  Week 12 (%) | -27.6 (25.10) | -50.9 (14.00) | -36.7 (24.07)
  Week 24 (%) | -37.4 (23.21) | -55.5 (12.62) | -44.5 (21.39)
  Week 52 (%) | -20.5 (36.95) | -52.8 (5.74) | -31.3 (33.69)

6. Secondary Outcome: Cardiopulmonary Exercise Testing (CPET) - Duration of Exercise
Description: Subjects performed maximal incremental exercise testing using an electronically braked upright cycle ergometer. Cycle ergometry is a method of CPET that may be feasible in subjects who have orthopedic, peripheral vascular, or neurological limitations that restrict weight bearing.
  Change from baseline to Week 25 and 52 as measured by the CPET Duration of Exercise (min)
Time Frame: Baseline, Week 25 and 52
Population: A subset of mITT subjects who were scheduled to perform CPET
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 10 | 5 | 15
Percent Change
  CPET Duration of Exercise Week 25 (min) | 0.8 (0.88) | 1.1 (1.43) | 0.9 (1.05)
  CPET Duration of Exercise Week 52 (min) | 0.6 (1.34) | 0.7 (1.46) | 0.6 (1.33)

7. Secondary Outcome: Cardiopulmonary Exercise Testing (CPET) - Peak Workload
Description: Subjects performed maximal incremental exercise testing using an electronically braked upright cycle ergometer. Cycle ergometry is a method of CPET that may be feasible in subjects who have orthopedic, peripheral vascular, or neurological limitations that restrict weight bearing.
  Percent change from baseline to Week 25 and 52 as measured by the CPET Peak workload (watt)
Time Frame: Baseline, Week 25 and 52
Population: A subset of mITT subjects who were scheduled to perform CPET
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 10 | 5 | 15
Percent Change
  Week 25 | 23.6 (20.87) | 38.4 (44.66) | 28.5 (30.04)
  Week 52 | 24.7 (26.17) | 13.0 (22.69) | 20.8 (24.90)

8. Secondary Outcome: Cardiopulmonary Exercise Testing (CPET) - O2 Pulse
Description: Subjects performed maximal incremental exercise testing using an electronically braked upright cycle ergometer. Cycle ergometry is a method of CPET that may be feasible in subjects who have orthopedic, peripheral vascular, or neurological limitations that restrict weight bearing.
  Percent change from baseline to Week 25 and 52 as measured by the CPET O2 pulse (ml/beat)
Time Frame: Baseline, Week 25 and 52
Population: A subset of mITT subjects who were scheduled to perform CPET
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 10 | 5 | 15
Percent Change
  Week 25 | 6.8 (14.17) | 13.5 (17.65) | 9.0 (15.13)
  Week 52 | 7.6 (27.89) | 2.0 (31.74) | 5.6 (28.22)

9. Secondary Outcome: Cardiopulmonary Exercise Testing (CPET) - Aerobic Efficiency
Description: Subjects performed maximal incremental exercise testing using an electronically braked upright cycle ergometer. Cycle ergometry is a method of CPET that may be feasible in subjects who have orthopedic, peripheral vascular, or neurological limitations that restrict weight bearing.
  Percent change from baseline to Week 25 and 52 as measured by the CPET Aerobic Efficiency (ml/watt).
  Note that decline in Aerobic Efficiency translate into an improvement
Time Frame: Baseline, Week 25 and 52
Population: A subset of mITT subjects who were scheduled to perform CPET
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 10 | 5 | 15
Percent Change
  Week 25 | -8.9 (15.41) | -6.0 (8.29) | -7.9 (13.02)
  Week 52 | -7.5 (28.39) | -9.8 (33.14) | -8.2 (28.52)

10. Secondary Outcome: Muscle Strength Testing (MST) - Knee Extension Test
Description: Change from baseline to Week 25 and 52 as measured by the peak force in MST knee extension test (newton meters).
Time Frame: Baseline, Week 25 and 52
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
Percent Change
  Week 25 | -0.6 (9.76) | 5.2 (7.63) | 1.7 (9.26)
  Week 52 | 3.3 (6.88) | 6.7 (8.87) | 4.7 (7.74)

11. Secondary Outcome: Muscle Strength Testing (MST) - Knee Flexion Test
Description: Percent change from baseline to Week 25 and 52 as measured by the peak force in MST knee flexion test (newton meters).
Time Frame: Baseline, Week 25 and 52
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
Percent Change
  Week 25 | -4.2 (24.83) | 9.4 (44.87) | 1.5 (34.39)
  Week 52 | -10.8 (22.72) | 8.2 (41.57) | -2.7 (32.69)

12. Secondary Outcome: Muscle Strength Testing (MST) - Elbow Flexion Test
Description: Percent change from baseline to Week 25 and 52 as measured by the peak force in MST elbow flexion test (newton meters).
Time Frame: Baseline, Week 25 and 52
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
Percent Change
  Week 25 | 12.0 (55.42) | 17.7 (41.82) | 14.1 (49.67)
  Week 52 | 49.7 (86.83) | 50.7 (59.81) | 50.1 (75.60)

13. Secondary Outcome: Adolescent Pediatric Pain Tool (APPT) - Pain Intensity
Description: The APPT is a validated, multidimensional tool to evaluate pain in children, adolescents, and young adults. The complete APPT is measured in three parts - Part 1 of the APPT scale determines the subject's pain locations using a body template. Part 2 of the APPT scale determines the intensity of the pain using a 10 cm visual analog scale (VAS) with the lowest point of the scale (0) labeled No Pain and the highest point on the scale (10) labeled Worst Possible Pain. Intermediate regions of the sale were labeled with 3 intermediate descriptors (Little Pain, Medium Pain, and Large Pain). Part 3 of the APPT scale characterizes the pain by tracking the number and percentage of words selected by subjects to describe their pain from a total of 57 choices. Part 2 corresponds most closely to other typically used pain scales (based on VAS) and for this reason the results from Part 2 are presented here.
  Change from baseline to Week 12, 24, and 52 in pain intensity.
Time Frame: Baseline, Week 12, 24, and 52
Population: Modified Intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week | All Subjects
Number analyzed (Participants) | 15 | 10 | 25
units on a scale
  APPT Word Graphic Rating Scale Week 12 | -2.3 (3.37) | -1.2 (2.23) | -1.8 (2.93)
  APPT Word Graphic Rating Scale Week 24 | -2.2 (3.68) | -1.2 (2.87) | -1.8 (3.33)
  APPT Word Graphic Rating Scale Week 52 | -0.8 (3.41) | -0.8 (3.04) | -0.8 (3.17)

ADVERSE EVENTS:
Time Frame: Study Period, up to 192 weeks or ETV
Description: All Adverse Events
Arm/Group | BMN 110 Weekly at 2.0 mg/kg/Week | BMN 110 Weekly at 4.0 mg/kg/Week
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/10
Other Adverse Events (participants affected / at risk) | 15/15 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 110 Weekly at 2.0 mg/kg/Week (N=15) | BMN 110 Weekly at 4.0 mg/kg/Week (N=10)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Enuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 110 Weekly at 2.0 mg/kg/Week (N=15) | BMN 110 Weekly at 4.0 mg/kg/Week (N=10)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Pectus carinatum (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (3) | 2 (2)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (2) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (18) | 3 (23)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (8) | 4 (11)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (21) | 4 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (33) | 5 (6)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (34) | 5 (10)
Catheter site pain (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (12) | 2 (5)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Infusion site bruising (General disorders) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 3 (6) | 2 (4)
Infusion site swelling (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 2 (3) | 0 (0)
Local swelling (General disorders) | 2 (3) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 9 (24) | 3 (9)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 2 (3) | 0 (0)
Enterobiasis (Infections and infestations) | 1 (3) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 3 (5)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (10) | 7 (16)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (5) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (13) | 5 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Inadequate analgesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 5 (8) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (28) | 5 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (13) | 1 (1)
Elbow deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (22) | 4 (5)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (8) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (89) | 7 (44)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (3)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Phobia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 4 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 4 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 4 (9) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (11) | 0 (0)
Catheterisation venous (Surgical and medical procedures) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Medical device removal (Surgical and medical procedures) | 0 (0) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish any data prior to multi-centre publication. If publication related to sub-sets of data it shall make reference to the relevant multi-centre publication. PI agrees to submit material to Sponsor for review up to 60 days prior to publication and incorporate all reasonable comments. During review, Sponsor may request that publication be delayed for up to 6 months from date of first submission to Sponsor in order for Sponsor to take steps to protect its proprietary information.